CLINICAL TRIAL: NCT01043406
Title: Safety and Effectiveness of a Seizure Advisory System in Epilepsy: A Feasibility Study (Victoria)
Brief Title: Seizure Advisory System Feasibility Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor restructuring.
Sponsor: NeuroVista Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVC1001
Record Dates: First submitted 2010-01-04; First posted 2010-01-06 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Epilepsy
Keywords: Epilepsy; Seizures; Advisory; Prediction
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm, Device Implant (Experimental)
  Interventions: Device: Seizure Advisory System

INTERVENTIONS:
Device: Seizure Advisory System — Implant of Seizure Advisory System followed by data collection for algorithm training and subsequent enabling of seizure advisory indicators.

SUMMARY:
The purpose of this prospective, single-arm, unblinded, multicenter clinical study is to evaluate the safety and effectiveness of the NeuroVista Seizure Advisory System (SAS) in patients with medically refractory epilepsy. A total of 15 subjects will be implanted at up to three study sites.

DETAILED DESCRIPTION:
This research project aims to evaluate the effectiveness of the SAS based on how well it provides subjects with signals (or "advisories") that they can see and hear to predict their "likelihood" of having a seizure. It does this by monitoring signals in the brain. A secondary purpose of the study is to learn whether the advisories improve subject quality of life or that of their caregiver.

The SAS is made up of three main components that work together to monitor the subject's brain signals and then relay their information to the subject: the leads, the implantable telemetry unit (ITU), and the personal advisory device (PAD). The leads will be placed on different areas of the subject's brain to record electrical signals. The leads are tunneled down the neck to an ITU that is implanted in the chest, similar to a pacemaker. The ITU wirelessly transmits information to the PAD, which is carried like a pager. It records and processes brain signals and may be able to advise subjects when a seizure is likely or unlikely to occur.

Following implantation with the SAS, subjects will return for five study visits for neurological examinations and quality of life assessments. Throughout the study, subjects must maintain their SAS; which includes daily recharging and data card replacement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has disabling partial seizures and/or secondarily generalized partial seizures. Disabling refers to seizures that are severe enough to cause injuries or to significantly impair areas of function such as employment, psychological or social wellbeing, or mobility.
2. Subject has failed treatment with a minimum of two AED's used in typical therapeutic dosages.
3. For three months prior to enrollment, subject's anti-epileptic medication dosages have been stable and subject has had at least two disabling seizures per month, on average, with a seizure-free interval not to exceed 45 days. Seizures must be separated by a minimum of eight hours not to be considered part of a cluster. A cluster, for the purpose of this criterion, shall be considered a single seizure.

Exclusion Criteria:

1. For three months prior to enrollment, subject's anti-epileptic medication dosages have not been stable, or subject has had more than 12 disabling seizures per month, on average, or there was a seizure-free interval longer than 45 days. Clinical seizures must be separated by a minimum of eight hours to not be considered part of a cluster. A cluster, for the purpose of this criterion, shall be considered a single seizure.
2. Subject is implanted with pacemaker, implantable cardiac defibrillator, cardiac management product, or a medical device that interferes with the SAS or with which the SAS interferes. This includes, but is not limited to, direct brain neurostimulators, spinal cord stimulators, vagus nerve stimulators (VNS), and cochlear implants. Patients with a vagus nerve stimulator implanted but turned off through the duration of the study may be enrolled, provided their clinical status has been stable for at least one month with VNS turned off.
3. Subject has been diagnosed with primary generalized seizures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The primary evaluation of safety will be an assessment of adverse events . | Adverse events through the primary safety endpoint four months post-implant.

SECONDARY OUTCOMES:
Seizure advisory performance will be assessed for the study population. | At the primary advisory performance endpoint at the conclusion of the Data Collection Phase (approximately 3 months post-implant) .
Clinical effectiveness will be evaluated. | At the primary clinical effectiveness endpoint 4 months following the commencement of the Advisory Phase (approximately 7 months post-implant)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Sheffield, VMD, PhD, Study Director — NeuroVista Corporation
Locations (3):
- Australia (3):
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St. Vincent's Hospital (Melbourne), Melbourne, Victoria
  - Austin Health, Melbourne, Victoria

REFERENCES:
- [Background] Snyder DE, Echauz J, Grimes DB, Litt B. The statistics of a practical seizure warning system. J Neural Eng. 2008 Dec;5(4):392-401. doi: 10.1088/1741-2560/5/4/004. Epub 2008 Sep 30. PMID 18827312
- [Derived] Cook MJ, O'Brien TJ, Berkovic SF, Murphy M, Morokoff A, Fabinyi G, D'Souza W, Yerra R, Archer J, Litewka L, Hosking S, Lightfoot P, Ruedebusch V, Sheffield WD, Snyder D, Leyde K, Himes D. Prediction of seizure likelihood with a long-term, implanted seizure advisory system in patients with drug-resistant epilepsy: a first-in-man study. Lancet Neurol. 2013 Jun;12(6):563-71. doi: 10.1016/S1474-4422(13)70075-9. Epub 2013 May 2. PMID 23642342